CLINICAL TRIAL: NCT07389811
Title: Effects of Telerehabilitation on the Occupational Performance of Stroke Patients Treated by an Occupational Therapy Service: a Randomized Clinical Trial
Brief Title: Telerehabilitation and Occupational Performance in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, André Tadeu Sugawara, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 86185525800000068
Record Dates: First submitted 2026-01-08; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Stroke
Keywords: Occupational Therapy; Telerehabilitation; Stroke; Public Health; Waiting Lists
MeSH Terms: conditions — Stroke | interventions — Telerehabilitation; Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation (Experimental): Participants in this group receive Occupational Therapy guidance via telehealth (telerehabilitation) focused on improving occupational performance.
  Interventions: Behavioral: Telerehabilitation in Occupational Therapy
- Waiting List (No Intervention): Participants allocated to this group remains on the waiting list for occupational therapy, following the natural course of functional improvement.

INTERVENTIONS:
Behavioral: Telerehabilitation in Occupational Therapy — Online guidance sessions for post-stroke patients and their caregivers, aimed at improving occupational performance, using standardized scales.
  Arms: Telerehabilitation

SUMMARY:
The objective of this randomized clinical trial is to evaluate the effects of using telerehabilitation (remote care) by occupational therapists on improving the performance and recovery of patients within the Brazilian Unified Health System (SUS) who have suffered a stroke and are on a waiting list for specialized rehabilitation care.

The main question it seeks to answer is:

* What are the effects of occupational therapy services provided through telerehabilitation for the population with stroke sequelae?
* Do the guidelines provided by telerehabilitation result in improved occupational performance (ability to perform activities of daily living) of the participants?

The researchers compare an experimental group (receiving telerehabilitation treatment) with a waitlist group (which will remain on the waitlist without receiving a specific intervention).

Participants are required to:

* Answer a sociodemographic questionnaire;
* Participate in assessments using standardized scales on basic and instrumental activities of daily living and use of the affected limb (Instrumental Activities of Daily Living Scale, Katz Scale, and Motor Activity Log).
* Receive and apply Occupational Therapy guidelines (if in the intervention group).

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable
* Diagnosis of sequelae of stroke (regardless of modified Rankin scale score)
* On a waiting list with medical indication for Occupational Therapy at IMREA HCFMUSP
* Access to a computer, tablet, or smartphone with internet connection allowing for video calls
* Ability to understand the Portuguese language
* Availability of a caregiver to assist during therapy sessions, if necessary

Exclusion Criteria:

* Clinically unstable patients (e.g., frail elderly with decompensated chronic diseases)
* High-risk pregnant women
* Lack of access to internet or devices required for telerehabilitation
* Absence of a caregiver when assistance is required for sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-07-27 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-26 (Actual)

PRIMARY OUTCOMES:
Change in "Katz Index of Independence in Activities of Daily Living" score indicating greater independence or dependence in performing basic activities of daily living after 2 months. | From enrollment to the end of treatment at 8 weeks
  The Katz Index (Brazilian version) assesses functional status in six activities: bathing, dressing, toileting, transferring, continence, and feeding. The total score ranges from 0 to 6. In this specific version, 0 indicates full independence (best outcome) and 6 indicates full dependence (worst outcome). Therefore, lower scores indicate a better outcome.
Change in "Lawton Instrumental Activities of Daily Living" score indicating greater independence or dependence in performing instrumental activities of daily living after 2 months. | From enrollment to the end of treatment at 8 weeks
  The Lawton Scale (Brazilian version) assesses independent living skills such as using the phone, shopping, food preparation, housekeeping, laundry, mode of transportation, responsibility for their own medications, and ability to handle finances. Scores range from 7 to 21. Higher scores indicate greater independence (better outcome).
Change in "Motor Activity Log" score for quantitative and qualitative analysis of the use of the affected upper limb. | From enrollment to the end of treatment at 8 weeks
  The MAL (Brazilian version) scale assesses how well the patient uses the affected upper limb. Participants rate the quality of movement on a scale from 0 (The weaker arm is not used) to 5 (Ability to use the weaker arm is just as good as before the stroke). The final score is the mean of the items. Higher scores indicate better movement quality (better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Physical Medicine and Rehabilitation of the Hospital das Clínicas of the Faculty of Medicine of USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
There will be no sharing of Individual Participant Data (IPD). This decision is based on Law Nº. 13.709, of August 14, 2018 (General Law on the Protection of Personal Data - LGPD), specifically regarding the protection of sensitive data (Article 5, item II), relating to health and sex life, genetics or biometrics. The disclosure of raw data, even if pseudonymized, may pose risks of re-identification of participants, who are vulnerable patients (post-stroke) treated by the Unified Health System (SUS) at IMREA FMUSP. The publication of results will occur exclusively in an aggregated and statistical manner, preserving medical confidentiality and the identity of volunteers, as recommended by the resolutions of the National Health Council (CNS/CONEP).

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-21): https://cdn.clinicaltrials.gov/large-docs/11/NCT07389811/Prot_SAP_ICF_000.pdf